CLINICAL TRIAL: NCT00836667
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Sertraline Hydrochloride 100 mg Tablets and Zoloft® 100 mg Tablets Administered as 1 x 100 mg Tablet in Healthy Subjects Under Fed Conditions.
Brief Title: Sertraline Hydrochloride 100 mg Tablets, Fed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 02071
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Sertraline hydrochloride 100 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Zoloft® 100 mg Tablets

INTERVENTIONS:
Drug: Zoloft® 100 mg Tablets — 1 x 100 mg, single-dose fed
  Arms: 2
Drug: Sertraline hydrochloride 100 mg Tablets — 1 x 100 mg, single-dose fed
  Arms: 1

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of sertraline hydrochloride 100 mg tablets (test) versus Zoloft® (reference) administered as 1 x 100 mg tablet under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be females and/or males, non-smokers, 18 years of age and older. Female subjects will be post-menopausal or surgically sterilized.
* Post-menopausal status is defined as absence of menses for the past 12 months.
* Sterile status is defined as hysterectomy, bilateral oophorectomy or tubal ligation at least 6 months ago.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical sub-investigator, would preven the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHG, or diastolic blood pressure lower than 50 or over 90 mmHg; or heart rate less than 50 or over 100 bpm) at screening.
* Subjects with BMI ≥ 30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%)
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical sub-investigator, contraindicates the subject's participation in this study.
* History of allergic reactions to sertraline or other related drugs (e.g. fluoxetine hydrochloride, fluvoxamine hydrochloride, paroxetine hydrochloride).
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine), use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural products, vitamins, garlic as supplement and products containing dextromethorphan) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows: less than 300 mL of whole blood within 30 days or; 300 mL to 500 mL of whole blood within 45 days or; more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have consumed food or beverages containing grapefruit (3.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* Past history of bipolar affective disorder or other active psychiatric diagnosis.
* History of seizures.
* Subjects with a clinically significant history of renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Intolerance to venipuncture.
* Breast-feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-03; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada